CLINICAL TRIAL: NCT05930626
Title: Biomarkers of Acrylamide, Glycidol, POPs, PFAS and Disease Outcomes and OMICs Signatures
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: The Swedish Research Council (Other Government)
Responsible Party: Principal Investigator, Agneta Åkesson, Professor, Karolinska Institutet
Other Study IDs: EXP-21-CV8301-OMICS
Record Dates: First submitted 2023-06-09; First posted 2023-07-05 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Disease; Cardiovascular Diseases; Cancer; Environmental Exposure
MeSH Terms: conditions — Disease; Cardiovascular Diseases; Neoplasms | interventions — glycidol; phosphoribosylformylglycinamidine synthetase

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SMC-C: Swedish Mammography Cohort-clinical (SMC-C) is a clinical sub-cohort established between 2003 and 2008, consisting of 5022 women, 56-80 years of age, living in Uppsala. These women have completed a detailed questionnaire on diet and lifestyle factors and underwent a health examination, dual-energy X-ray absorptiometry and biological sampling.
  Interventions: Other: Biomarkers of acrylamide, glycidol, POPs, PFAS
- 60YO: The cohort of 60-years olds (60YO) was established with the aim to study CVD etiology and consists of 4,232 men and women aged 60 years who were randomly selected from Stockholm County and with baseline examination during 1 year in 1997-98. The study participants underwent a health examination, completed a questionnaire, and donated blood samples.
  Interventions: Other: Biomarkers of acrylamide, glycidol, POPs, PFAS

INTERVENTIONS:
Other: Biomarkers of acrylamide, glycidol, POPs, PFAS — These are food contaminants (acrylamide, glycidol) and environmental pollutants (POPs, PFAS). Assess the associations between biomarkers of acrylamide and glycidol exposure and disease outcomes in a case-cohort study based on two prospective cohorts with biobanks. The investigators also aim to assess the exposure-affected OMICS signatures and molecular pathways underlying disease development (specifically cardiovascular diseases such as myocardial infarction and stroke and cancer such as breast-, endometrial and colorectal cancer) for these exposures along with POPs and PFAS using a prospective cohort study utilizing and integrating various 'OMICs' technologies.

SUMMARY:
The aim of the project is to assess the associations between biomarkers of acrylamide and glycidol exposure and disease outcomes in a case-cohort study based on two prospective cohorts with biobanks. The investigators also aim to assess the exposure-affected OMICS signatures and molecular pathways underlying disease development (specifically cardiovascular diseases such as myocardial infarction and stroke and cancer such as breast-, endometrial and colorectal cancer) for these exposures along with persistent organic pollutants (POPs) and per- and polyflouroalkyl substances (PFAS) using a prospective cohort study utilizing and integrating various 'OMICs' technologies.

ELIGIBILITY:
Inclusion Criteria:

* 60YO: Men and women of 60 years old residing in Stockholm
* SMC-C: Women residing in Uppsala

Exclusion Criteria:

* Subjects will be excluded if they had the outcome under investigation at baseline

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 60YO: Men and women of 60 years of age living in Stockholm SMC-C: Women living in Uppsala
Sampling Method: Probability Sample
Enrollment: 9254 (Actual)
Dates: Start 1997-01-01 (Actual); Primary Completion 2008-12-31 (Actual); Study Completion 2008-12-31 (Actual)

PRIMARY OUTCOMES:
Cardiovascular disease | From baseline beginning in 2003 through 2017
  Using International Classification of Diseases (ICD) codes to assess cardiovascular disease (CVD) incidence (myocardial infarction and stroke, ICD10: I21 and I63)
Cancer | From baseline (2003 for SMC-C and 1997 for 60YO) until the latest available follow-up, currently 2021
  Using ICD codes to assess cancer (such as ICD-10: C18, C20, C50, C54)

IPD SHARING:
Plan to Share IPD: No
Individual participant data is available from registers at Statistics Sweden and National Board of Health and Welfare in Sweden.